CLINICAL TRIAL: NCT07111663
Title: An Observational Study of Individuals With Isolated Dystonia
Status: Recruiting | Type: Observational
Sponsor: Vima Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: VIM0423-401
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Isolated/Primary Dystonia That Affects More Than One Region of the Body
Keywords: Dystonia, Isolated Dystonia, Primary Dystonia, Cervical Dystonia
MeSH Terms: conditions — Dystonia; Dystonic Disorders; Torticollis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Isolated (or Primary) Dystonia Cohort: This is a single-arm noninterventional, prospective observational study enrolling up to 200 male and female participants (ages 12 - 65 years, inclusive) that have been diagnosed with isolated dystonia for at least one year prior to the first study visit. Candidates with focal dystonia (i.e., only one body part affected) are not eligible for participation. However, the Investigator may query such patients to determine if symptoms have spread to other regions, which may allow them to be eligible for study entry.

SUMMARY:
This is an observational study in individuals with isolated (or primary) dystonia that involves more than one body region. The purpose of the study is to collect detailed information to help your physician and other researchers understand how dystonia impacts your and other patients' lives and how the disease changes over time. The study may also help researchers better understand the clinical scales that are commonly used to evaluate dystonia symptoms and how they affect various areas of life such as well-being, pain, relationships and social interactions, and progress over time. Because this is an observational study, you will not receive any interventional treatment in the study.

DETAILED DESCRIPTION:
The primary goal of this observational study is to further characterize and quantify disease severity and impact (including change over time) in individuals with either segmental, multifocal, or generalized dystonia in a structured manner, utilizing and comparing various well-known scales. In addition, medication history and any intercurrent events related to the participant's health (such as, but not limited to, hospitalizations, new diagnoses, etc.) will be captured. This study will provide standardized data to support planned future interventional clinical studies in this patient population and will provide a greater understanding of the population under study and the performance of clinical ratings scales.

ELIGIBILITY:
Inclusion Criteria: Each participant must meet the following criteria at Visit 1 to be eligible to continue in the study:

* The participant is willing to sign an informed consent form indicating that he/she understands the purpose of the study; understands and can perform, complete, and comply with all the assessments that are required during the study; and is willing to participate in the study.
* The participant is a male or female between 12 and 65 years of age (inclusive).
* The participant has a clinical diagnosis of isolated (or primary) dystonia for at least one year prior to Visit 1 and meets the study definition of segmental/multifocal or generalized dystonia at Visit 1.

Exclusion Criteria: Any participant who meets any of the following criteria at Visit 1 will be excluded from this study:

* The participant has a diagnosis of focal dystonia at Visit 1.
* The participant has a diagnosis of dopa-responsive dystonia, secondary dystonia, or psychogenic/functional dystonia.
* The participant has any significant ongoing disease, disorder, laboratory abnormalities, alcohol or illicit drug abuse or dependence, environmental factor, or any ongoing or history of any medical or surgical condition that in the judgment of the investigator, in consultation with the medical monitor and/or sponsor's designee, might jeopardize the participant's safety, impact the scientific objectives of the clinical study, or interfere with participation in the clinical study.
* The participant has a history of any psychiatric or cognitive impairment disorder that, in the opinion of the investigator, may interfere with study conduct.
* The participant has had myotomy or denervation surgery in any affected muscles (e.g., peripheral denervation and/or spinal cord stimulation).
* The participant has marked limitation on passive range of motion that suggests contractures or other structural abnormality (e.g., cervical contractures or cervical spine syndrome).
* The participant has undergone deep brain stimulation (DBS) surgery (even if implant deactivated).

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Isolated (Primary) Dystonia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Burke-Fahn-Marsden (BFM) Dystonia Rating Scale | From start of treatment through 4 months
  The BFM was developed to quantitatively assess primary dystonias (Burke 1985). It is composed of 2 subscales: a movement subscale, based on the clinician's evaluation of the patient in nine body areas, and a disability subscale, based on the participant's report of disability in activities of daily living.

SECONDARY OUTCOMES:
Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS-2) | From start of treatment through 4 months
  The TWSTRS-2 scale is used to assess cervical dystonia. It includes 3 subscales that evaluate symptom severity, disability, and pain. The severity scale is clinician-rated and the disability scale is patient-rated based on 6 items related to work, activities of daily living, driving, reading, watching TV, and outside activities.
Clinical Global Impression of Severity (CGI-S) | From start of treatment through 4 months
  The CGI-S score is used by the Investigator to determine, in a global sense, how severe the patients' blepharospasm is in the context of other blepharospasm patients. Increased scores indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Vima Site #004, Scottsdale, Arizona
  - Vima Site #028, Sun City, Arizona
  - Vima Site #010, Aliso Viejo, California
  - Vima Site #030, Los Angeles, California
  - Vima Site #022, Palo Alto, California
  - Vima Site #019, Englewood, Colorado
  - Vima Site #003, Boca Raton, Florida
  - Vima Site #009, Gainesville, Florida
  - Vima Site #008, Miami, Florida
  - Vima Site #031, Orlando, Florida
  - Vima Site #005, Atlanta, Georgia
  - Vima Site #027, Chicago, Illinois
  - Vima Site #007, Olney, Maryland
  - Vima Site #002, Farmington Hills, Michigan
  - Vima Site #014, Albuquerque, New Mexico
  - Vima Site #017, Commack, New York
  - Vima Site #018, New York, New York
  - Vima Site #024, New York, New York
  - Vima Site #029, Portland, Oregon
  - Vima Site #020, Philadelphia, Pennsylvania
  - Vima Site #021, Charleston, South Carolina
  - Vima Site #016, Memphis, Tennessee
  - Vima Site #006, Nashville, Tennessee
  - Vima Site #025, Dallas, Texas
  - Vima Site #026, Georgetown, Texas
  - Vima Site #012, Houston, Texas
  - Vima Site #011, Richmond, Virginia
  - Vima Site #023, Kirkland, Washington
  - Vima Site #015, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No